CLINICAL TRIAL: NCT02842190
Title: Nasal Intermittent Positive Pressure Ventilation Versus Bi-level Nasal Continuous Positive Airway Pressure Following Extubation in Infants ≤ 1250 g Birthweight
Brief Title: NIPPV Versus Bi-level Nasal Continuous Positive Airway Pressure Following Extubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, nilüfer okur, NEONATOLOGY, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NIPPV-2016
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Intubation Complication; PreTerm Birth
Keywords: Neonatal; NIPPV; BIPAP; Extubation failure
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIPPV (Active Comparator): NIPPV after ekstubation
  Interventions: Device: NIPPV
- BIPAP (No Intervention): BIPAP after ekstubation

INTERVENTIONS:
Device: NIPPV — after ekstubation
  Arms: NIPPV

SUMMARY:
Mechanical ventilation is important in the care of preterm infants with respiratory failure, but may be associated with lung injury. Efforts are needed to avoid or minimize the use of mechanical ventilation. However, there is no consensus on the best non-invasive ventilation mode after extubation in preterm infants.

Objective: To compare the effectiveness of nasal intermittent positive pressure ventilation (NIPPV) versus bi-level nasal continuous positive airway pressure (BIPAP) following extubation in preterm infants ≤ 1250 g birthweight.

DETAILED DESCRIPTION:
In this study , mechanically ventilated preterm infants with birthweight ≤1250 g will screen for eligibility. Infants with major congenital malformations, neuromuscular disease and lack of parental consent were excluded. Enrolled infants will randomize into two study groups (NIPPV group and BIPAP group) following the decision to extubate by using sealed opaque envelopes. Extubation criteria are; loaded with caffeine according to standard clinical protocol, satisfactory blood gases (pH of more than 7.25), mean airway pressure of 7 cm water or less, fractional inspired oxygen concentration of 35 % or less and good respiratory effort.

Non-invasive respiratory support will deliver using the device of SLE 5000 (Specialised Laboratory Equipment, South Croydon, United Kingdom) in NIPPV group and infant flow- deriver device (Viasys Corp, Care Fusion, CA) in BIPAP group. The short binasal prongs will use as interface. The initial ventilator parameters for NIPPV were: PIP levels set 2 cm H2O above the pre-extubation PIP, PEEP: 5 cm H2O, rate the same as was being given before extubation and for BiPAP were: lower CPAP levels 4 to 6 cmH2O (maximum 7 cmH2O) and higher CPAP levels 8 to 9 cmH2O (maximum 10 cmH2O), Thigh 0.5-0.6 second, and a pressure exchange rate of 20-30/ minute, with the lowest adjusted FiO2 to maintain an oxygen saturation of 90% to 95%.

Extubation failure was defined as: development of respiratory acidosis (blood gases with pH < 7.2 and PaCO2> 60 mmHg), or hypoxemia (blood gases with PaO2 < 50 mmHg despite oxygen supplementation of 60 percent), or severe apnea requiring mask ventilation.

Surfactant requirement is goingto evaluate in all infants after NICU admission. Poractant alfa was administered if necessary.

The primary end-point, rate of extubation failure within 96 hours following first extubation, will compared between the groups. Short and long-term neonatal outcomes will also evaluate.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated preterm infants with birthweight ≤1250 g

Exclusion Criteria:.

* Infants with major congenital malformations, neuromuscular disease and lack of parental consent

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2016-01-15; Primary Completion 2017-06-30 (Actual); Study Completion 2019-10-15 (Estimated)

PRIMARY OUTCOMES:
Rate of extubation failure | within 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Serife Suna Oguz, Study Director — Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey. Recruiting; Nurdan Uras, Study Chair — Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey. Recruiting
Locations (1):
- Zekai Tahir Burak Maternity Teaching hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Okur N, Buyuktiryaki M, Sari FN, Dizdar EA, Oguz SS. Ventilator-delivered nasal intermittent positive pressure ventilation versus nasal biphasic positive airway pressure following extubation in infants </=1250 g birth weight: a randomized trial. J Matern Fetal Neonatal Med. 2022 Feb;35(4):752-758. doi: 10.1080/14767058.2020.1731462. Epub 2020 Feb 27. PMID 32106721